CLINICAL TRIAL: NCT02909725
Title: The Blossom Project: "BlossomUP" Evaluating Methods to Decrease Sedentary Time in Pregnancy
Brief Title: The Blossom Project: "BlossomUP" Methods to Decrease Sedentary Time in Pregnancy
Acronym: BUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Christina Campbell, Associate Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #15-749
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Sedentary Lifestyle; Diabetes Mellitus, Gestational
Keywords: Physical activity; Sedentary time; Pregnancy; Pregnant women; Weight gain
MeSH Terms: conditions — Sedentary Behavior; Diabetes, Gestational; Motor Activity; Weight Gain | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Limit accumulation of sedentary time (Experimental): Group 1 (SR): Participants will be asked to limit the accumulation of prolonged bouts ( >50 minutes) of sedentary time.
  Interventions: Other: Limit accumulation of sedentary time
- Walk 30 minutes most days of the week (Experimental): Group 2 (WALK): Participants will be asked to walk 30 minutes per day on most days of the week.
  Interventions: Other: Walk
- Normal daily routine; Usual Care (Active Comparator): Group 3 (UC): Participants will be asked to continue on with their normal daily routine. The usual care group will receive no form of intervention.
  Interventions: Other: Normal daily routine; Usual Care

INTERVENTIONS:
Other: Limit accumulation of sedentary time — Participants in this group receive a Fitbit Alta activity monitor, worn on the wrist for the entire intervention. The Alta is a fitness tracker designed to help individuals track their sedentary and physical activity behaviors when paired with an external device (e.g. iPhone, computer). The Sensewear armband and ActivPAL are not worn as part of the intervention; they are assessment tools used at the beginning and end of the study.
  Each participant will have a Fitbit account set up with a Blossom Project username code to ensure privacy of the participant's identity. Participants will be asked to achieve a goal of 250 steps/hour. Using the "reminder to move" function, if a participant has not reached the hourly goal at 50 minutes, the Alta will vibrate, cueing the participant to walk.
  Arms: Limit accumulation of sedentary time
Other: Walk — Participants in this group receive a Fitbit Charge activity monitor. There is no "reminder to move" function on this band. The Charge, worn on the wrist for the entire intervention is a fitness tracker designed to help individuals track their physical activity when paired with an external device. The Sensewear armband and ActivPAL are not worn as part of the intervention; they are assessment tools used at the beginning and end of the study.
  Each participant will have a Fitbit account set up with a Blossom Project username code to ensure privacy of the participant's identity. Participants will be asked to meet current pregnancy physical activity recommendations; walking 30 minutes, most days of the week (150 minutes/week). Participants can use the app to view their "active minutes."
  Arms: Walk 30 minutes most days of the week
Other: Normal daily routine; Usual Care — Participants in this group will not be provided with a Fitbit Charge activity monitor, as participants will be asked to simply continue on with their normal daily routine. The Sensewear armband and ActivPAL are not worn as part of the intervention; they are assessment tools used at the beginning and end of the study.
  Arms: Normal daily routine; Usual Care

SUMMARY:
Multiple studies have demonstrated a very low prevalence of women meeting physical activity and weight gain recommendations during pregnancy. Additionally, previous Blossom Project studies have shown that when pregnant women engage in a 20 minute walk each day, they spend significantly more time sitting in addition to longer bouts of sitting resulting in increased total sedentary time. We are going to test which method works best to decrease sitting time, and how those methods effect metabolic parameters such as insulin resistance and blood glucose. This study will consist of three groups, each utilizing a commercially available fitness tracker, Fitbit. Group 1 (SR): will reduce sedentary time by interrupting prolonged sitting. Group 2 (WALK): will reduce sedentary time via walking. Group 3 (UC): will continue on with their normal daily routine; usual care.

DETAILED DESCRIPTION:
Pregnant women will be recruited using mass email recruitment, fliers posted at local community settings, and at local OBGYN offices in Ames, IA. Pregnant women will be recruited between 16 and 22 weeks gestation. Interested individuals will contact the Blossom Project staff for further information.

A randomized controlled design will be used. Following baseline data collection, women will be randomized into group 1 (n=12), group 2 (n=12) or group 3 (n=12).

For this study, the goal is to have a total of 10 women in each of the three groups. With an attrition rate of 15%, investigators plan to enroll a total of 36 women. Furthermore, increased enrollment numbers will cover inconsistencies that may arise with missing or uninterpretable data.

Individuals who contact the Blossom Project will be screened for eligibility. Individuals that meet the inclusion and exclusion criteria will meet with a Blossom Project staff member to sign an informed consent form approved by the Iowa State University Institutional Review Board (ISU-IRB). A "medical consent form" (not the consent form for the study participant) will be sent to the woman's primary obstetric provider asking to confirm qualification criteria. Participants will then be asked to complete a medical history questionnaire.

Eligible participants will be asked to participate in a 6 week intervention. Participants will report to the Nutrition Wellness Research Center (NWRC) either on campus (HNSB 2021, 2022, 2023) or the facility located at 2325 North Loop Drive, Suite 6100, Ames, Iowa 50010 at the start of week 1 and week 6. Week 1 and 6 include an 8-day data collection period outlined below. Weeks 2-6 include the intervention period.

Data that will be collected during each of the data collection periods will include:

Week 1 Visit: Pregnant between 16 and 22 weeks of gestation:

* Consent form: Participants will meet with a staff member to discuss the consent form and requirements of the study. Signed informed consent will be obtained from each participant.
* Medical provider consent: Medical providers will confirm qualification criteria for each participant. The medical provider consent must be received prior to a woman beginning participation in the study. Participants will sign this form at visit 1 to grant Blossom Project staff the permission to contact their medical provider.
* Medical history questionnaire: Each participant will fill out a medical history questionnaire.
* Physical activity assessment: Participants will receive verbal and written instructions on how to collect data regarding their physical activity. Each participant will wear 2 activity monitors to assess physical activity patterns over the 8-day monitoring period during baseline data collection and the sixth week of the study. The sensors will be worn on the left arm over the triceps muscle (SenseWear Mini armband) and on the right leg over the quadriceps muscle (activPAL). All of these monitors have been used in our previous pregnancy studies with minimal complaints. Participants are required to record all their daily activities in a physical activity log that will be provided. The log is required to be recorded over the same consecutive 8 days for 24 hours a day that the 2 activity monitors are worn.
* Dietary assessment: Participants will receive verbal instructions on how to collect data regarding their dietary intake. Each woman will complete a 3-day weighed diet record which requires her to weigh and record all food and beverages consumed for 2 weekdays and 1 weekend day. Detailed written instructions will also be provided in a binder in a data collection bag with a dietary scale.

  * Anthropometric measurements: Height and weight will be measured.
  * Scheduling of follow-up appointment: Participants will schedule a time to return to the research facility the following week to return all monitors and materials (diet record, data collection bag, dietary scale).

Week 6 Visit: Between 24-28 weeks gestation:

* Physical activity assessment via two monitors: SenseWear armband and the activPAL
* 3-day weighted diet record
* Anthropometric measurements: Weight and 2-hour Oral Glucose Tolerance Test: The oral glucose tolerance test will consist of providing a fasted blood sample (following an overnight fast of 10-12 hours), consuming a 75-gram oral glucose solution and a blood sample at 60 minutes and 120 minutes following the consumption of the glucose solution. During this 2-hour period, the participant will be asked to remain seated at the research facility. The blood draw will be conducted by an experienced phlebotomist.

In order to protect the privacy of participants within the study records identifying participants will be kept confidential to the extent allowed by applicable laws and regulations. Records will not be made publicly available. To ensure confidentiality to the extent allowed by law, the following measures will be taken. Participants will be assigned a unique code that will be used on forms instead of their name. The signed consent form, medical provider consent form, and release of medical information forms will all need the woman's full name to identify her to her prenatal clinic and delivering hospital. These forms will be locked in a separate filing cabinet from the forms with the participant codes to prevent identification of the participants. If the results are published, the identity will remain confidential. The data obtained from the study will be regarded as privileged and confidential. The privacy will be maintained in any future analysis and/or presentation of the data with the use of coded identifications for each participant's data. Only members of the Blossom Project lab staff will have access to the data and study records. All data will be stored in a locked file cabinet with access only by the principal investigator and project staff. This data will be kept on hand in a separate locked file in the PI's laboratory (HNSB 1109, Iowa State University) until the results of the study have been published. Identifiers will be kept separate from the data. All electronic data is stored on a shared drive only accessible to the principal investigator and project staff which requires a password to access.

For statistical analysis data we will be comparing sitting time (total and bouts of 30 and 60+ minutes) and walking time (total and bouts of 10, 20 and 30+ minutes) between groups. Group differences will be assessed using analysis of variance with post-hoc bonferonni for significant differences. Where appropriate, analyses will adjust for potentially important covariates. Relationships between sitting time, walking time and rate of weight gain will be evaluated. Responses will be transformed when necessary. Statistical significance will be set at p < 0.05 and adjusted for any multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant with one fetus between 16 and 22 weeks of gestation
* Receiving regular prenatal care, and physician documented approval to participate in this study
* Only inactive women will be enrolled; "inactive" is defined as self-reported participation in less than 3 planned exercise sessions/week for < 30 minutes per day for at least 6 months prior to conception.

Exclusion Criteria:

* History of smoking during pregnancy;
* History of the following chronic diseases: Type 1 diabetes, cardiovascular disease or renal disease
* Pre-pregnancy BMI > 40 kg/m2;
* Inability to communicate due to language barrier or mental status;
* Not having access to an UpBand compatible mobile device;
* Any adverse reactions to armband monitors (e.g. metal allergies, electromagnetic devices)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Time Spent Sedentary | From baseline to final data collection (week 6)
  Change in time spent sedentary as measured by data collected via ActivPAL analysis.

SECONDARY OUTCOMES:
Maternal Insulin Resistance | Maternal 24th-28th week of gestation
  Plasma glucose concentrations and insulin resistance as measured from a oral glucose tolerance test.

OTHER OUTCOMES:
Maternal Body Weight Change | From baseline to final data collection (week 6)
  Gestational weight gain as measured by final data collection (week 6) weight minus self-reported pre-pregnancy weight.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Campbell, PhD, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No